CLINICAL TRIAL: NCT04823858
Title: A Prospective Data Collection Study of Patients Treated With a Single-Level Lumbar Interbody Fusion Stabilized With Pedicle Screws
Brief Title: 3Spine Lumbar Fusion Real World Evidence Study
Status: Active, not recruiting | Type: Observational
Sponsor: 3Spine (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: 3Spine Lumbar Fusion Study
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Lumbar Spine Degeneration
Keywords: Posterior lumbar interbody fusion; Transforaminal lumbar interbody fusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Examination Group: There will only be one arm of subjects in this study. The arm will include subjects who plan to undergo a single-level TLIF/PLIF stabilized with pedicle screws and meet all of the eligibility criteria.
  Interventions: Procedure: Lumbar Interbody Fusion

INTERVENTIONS:
Procedure: Lumbar Interbody Fusion — The TLIF/PLIF system includes a TLIF/PLIF interbody cage and a pedicle screw system (4 screws with 2 rods). Any FDA cleared TLIF/PLIF interbody cage and pedicle screw system is acceptable for this study (with the exception of PEEK rods) as long as it is implanted per the package insert. No subjects implanted with an off-label use of a device are permitted for this study.

SUMMARY:
This study is designed to collect real world evidence (RWE) safety and efficacy data on patients who plan to undergo a single-level Transforaminal lumbar interbody fusion (TLIF) or Posterior lumbar interbody fusion (PLIF) instrumented with pedicle screws, using the framework of a prospective clinical study (with defined enrollment criteria and pre-specified research follow-up timepoints).

DETAILED DESCRIPTION:
A prospective, multi-center (up to 25), non-blinded study of patients who plan to undergo a single-level Transforaminal lumbar interbody fusion (TLIF) or Posterior lumbar interbody fusion (PLIF) stabilized with pedicle screws. Investigators will only select those patients who are planned for treatment with on-label use of FDA cleared TLIF/PLIF devices (cage and screw system).

At least 200 subjects with a potential sample size re-estimation at completion. The subjects will return for follow-up at 6-weeks, 3-months, 6-months, and then annually for 5-years post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 21-80 (inclusive) with at least 3 years of life expectancy;
2. Subject plans to undergo a one-level Open or Mini-Open TLIF or PLIF procedure (stabilized with pedicle screws) independent of this research protocol;
3. Subject is to be treated with on-label use of an FDA-cleared TLIF or PLIF cage(s) and pedicle screw system independent of this research protocol;
4. The subject has a primary diagnosis of symptomatic lumbar degeneration with or without foraminal or recess stenosis of the lumbar spine at a single level from L1/L2 to L5/S1 confirmed by subject history and radiographic imaging (CT, MRI, X-rays) with no more than a Grade 1 (<25% translation) spondylolisthesis. Symptomatic lumbar degeneration that may be associated with a co-morbid condition such as:

   1. Herniated nucleus pulposus;
   2. Scarring/thickening of the ligamentum flavum, annulus fibrosus, or facet joint capsule;
   3. Facet joint degeneration/osteophyte formation;
   4. Spondylosis (defined by the presence of osteophytes);
   5. Disc degeneration and/or annular degeneration; and/or
   6. Lumbar stenosis defined by spinal cord or nerve root compression;
5. Exhausted conservative treatment (e.g. bed rest, physical therapy, medications, transcutaneous electrical nerve stimulation (TENS), manipulation, and/or spinal injections) for at least 3 months or has a neurologic emergency;
6. Preoperative Oswestry Disability Index score >/= 40/100 at baseline;
7. Psychosocially, mentally and physically able and willing to fully comply with this protocol including adhering to follow-up schedule and requirements and filling out forms; and
8. Signed informed consent.

Exclusion Criteria:

1. More than one vertebral level requiring treatment;
2. Previous instrumented surgery (i.e.: anterior disc replacement, spinal fusion, interspinous device, etc.) at the index lumbar level or an adjacent level;
3. Degenerative or lytic spondylolisthesis greater than Grade 1 (<25% translation);
4. Rotatory scoliosis at the level to be treated;
5. Congenital bony and/or spinal cord abnormalities at the level to be treated;
6. Subcaudal defect, disrupting the integrity of the pedicle;
7. Clinically compromised vertebral bodies at the involved level due to current or past trauma, e.g., by the radiographic appearance of the fracture callus, malunion or nonunion;
8. Disrupted anterior longitudinal ligament at the index level;
9. Overlying thoracolumbar kyphosis (greater than or equal to 15 degrees) within one level (includes target and adjacent level) of the level to be treated;
10. Back pain of unknown etiology without leg pain;
11. Severe spondylosis at the level to be treated as characterized by any of the following:

    1. Autofusion (solid arthrodesis) determined radiographically (CT);
    2. Totally collapsed disc, or;
    3. Vertebral body that cannot be mobilized;
12. Known allergy to cobalt, chromium, molybdenum, nickel, polyethylene, titanium, or vitamin E;
13. Unable to undergo a CT scan or other radiograph assessments;
14. Osteopenia: The SCORE/MORES will be utilized for all females age <50 and males age <55 to screen if a DEXA scan is indicated. If SCORE/MORES value ≥ 6, then a DEXA scan is required. A DEXA scan is indicated for all females age ≥50 and all males age ≥55. If DEXA is required, exclusion will be defined as a DEXA bone density measured T score ≤ -1. An existing DEXA is allowed if completed within 6 months of subject screening;
15. Has history of any endocrine or metabolic disorder known to affect osteogenesis (e.g.: Paget's disease, renal osteodystrophy, Ehler-Danlos syndrome, or osteogenesis imperfecta);
16. Insulin-dependent diabetes mellitus;
17. Lactating, pregnant or interested in becoming pregnant in the next 3 years;
18. Active infection - systemic or local;
19. Any medical condition requiring treatment with any drug known to potentially interfere with bone/soft tissue healing or receiving radiation therapy that is expected to continue for the duration of the study;
20. Body Mass Index > 40;
21. Recurrent history of deep vein thrombosis, symptoms of arterial insufficiency, or thromboembolic disease;
22. Systemic disease including Lupus disease, Reiter's disease, Rheumatoid disease, AIDS, HIV, hepatitis or autoimmune disease that requires immunosuppressive therapy, including biologics, for systemic inflammation;
23. Spinal tumor;
24. Active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years;
25. Any degenerative muscular or neurological condition that would interfere with evaluation of outcomes, including but not limited to Parkinson's disease, amyotrophic lateral sclerosis (ALS), or multiple sclerosis;
26. Has chronic or acute renal and/or hepatic impairment and/or failure or prior history of renal and/or hepatic parenchymal disease;
27. Has a Waddell Signs of Inorganic Behavior score of 3 or greater;
28. In the opinion of the investigator, the subject has a behavioral, cognitive, social or medical problem that may interfere with the assessment of the safety or effectiveness of the device;
29. Current or recent history of chemical/alcohol abuse or dependency using standard medical definition of Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) code;
30. Currently smoking or using tobacco products, including e-cigarette products (e.g., vaping); (Use within 30 days of surgery date is considered 'current');
31. Currently pursuing or in active spinal litigation for medical negligence, or trauma, or workers compensation;
32. Is a prisoner, incarcerated, or has been coerced to participate in the study that could impact the validity of results;
33. Is currently participating in an investigational therapy (device and/or pharmaceutical) within 30 days prior to entering the study or such treatment is planned during the 24 months following enrollment into the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects participating in this study will be recruited from the investigators' standard patient populations. Only patients who plan to undergo an Open or Mini-Open TLIF or PLIF procedure independent of this research protocol, are considered for study.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) Score | 24 months compared to baseline
  Improvement of at least 15 points in ODI score (out of 100). The ODI is a self-reported questionnaire that contains ten sections concerning intensity of pain, lifting, personal care, walking, sitting, sexual function, standing, social life, sleeping and traveling.
Neurological Status | 24 months compared to baseline
  Absence of deterioration in neurological status compared to baseline examinations. Neurological examination will consist of a motor and sensory examination at each in person study visit conducted per physician standard of care.
Secondary surgical intervention (SSI) | 24 months
  Subject success will be determined with the absence of a secondary surgical intervention including revision, re-operation, removal, or supplemental fixation at the index level.
Serious device-related adverse events (SDAE) | 24 months
  Subject success will be determined with the absence of any serious device-related adverse events (SDAE)

SECONDARY OUTCOMES:
Visual Analog Score (VAS) - Worst Leg | 24 months compared to baseline
  Improvement in VAS - Worst leg of 20mm at 24 months compared to baseline. The VAS is a measurement instrument that measures the amount of pain that a subject feels ranges across a continuum from none to an extreme amount of pain.
VAS - Back | 24 months compared to baseline
  Improvement in VAS - Back pain of 20mm at 24 months compared to baseline
ODI | 24 months compared to baseline
  Improvement in ODI of 15 points at 24 months compared to baseline
ODI | 24 months compared to baseline
  Mean change in ODI over time intervals
VAS | 24 months compared to baseline
  Mean change in leg VAS over time intervals
VAS | 24 months compared to baseline
  Mean change in back VAS over time intervals

OTHER OUTCOMES:
PROMIS scores (Physical Function) | 24 months relative to the baseline
  Improvement in PROMIS scores (PROMIS Physical Function) compared to baseline
PROMIS scores (Depression) | 24 months relative to the baseline
  Improvement in PROMIS scores (PROMIS Depression) compared to baseline
PROMIS scores (Anxiety) | 24 months relative to the baseline
  Improvement in PROMIS score (PROMIS Anxiety) compared to baseline
PROMIS scores (Social roles/activities) | 24 months relative to the baseline
  Improvement in PROMIS score (PROMIS Social Roles/activities) compared to baseline
Demographics | 24 months
  The study will examine the patient population through descriptive statistics of the demographic variable - age
Demographics | 24 months
  The study will examine the patient population through descriptive statistics of the demographic variable - Body Mass Index (BMI)
Demographics | 24 months
  The study will examine the patient population through descriptive statistics of the demographic variable - gender
Intra-Operative Variables | 24 months
  The study will examine the patient population through descriptive statistics of the intra-operative variable - surgery time.
Intra-Operative Variables | 24 months
  The study will examine the patient population through descriptive statistics of the intra-operative variable - blood loss
Time to first SSI | 24 months
  Time to first SSI including specific actions (removal, revision, replacement, supplemental fixation) at the index or adjacent level
Radiographic fusion | 24 months
  Radiographic fusion as defined by the Image Review Charter and assessed by an independent core laboratory.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Todd Lanman MD, Inc., Beverly Hills, California
  - University of Colorado, Aurora, Colorado
  - Steamboat Orthopedics and Spine Institute (SOSI), Steamboat Springs, Colorado
  - Spine & Orthopedic Center, Deerfield Beach, Florida
  - Florida Orthopaedic Institute, Temple Terrace, Florida
  - Strenge Spine Institute, Paducah, Kentucky
  - The Spine Center of Louisiana, Baton Rouge, Louisiana
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Upstate Orthopedics, East Syracuse, New York
  - NYU Langone, Spine Research Center, New York, New York
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Pinehurst Surgical Clinic, Pinehurst, North Carolina
  - Vertrae, Miamisburg, Ohio
  - OrthoNeuro, New Albany, Ohio
  - Oklahoma City Clinical Research Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Center for Sports Medicine and Orthopaedics, Chattanooga, Tennessee
  - Ortho San Antonio, San Antonio, Texas
  - The Disc Replacement Center, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: No